CLINICAL TRIAL: NCT04126811
Title: Single-center, Open, Non-randomized, Phase II Prospective Study of Apatinib Combined With Chemotherapy in the Treatment of Unresectable Soft Tissue Sarcoma
Brief Title: Apatinib Combined With Chemotherapy in the Treatment of Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2019145
Record Dates: First submitted 2019-09-30; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; apatinib; Jilong Yang
MeSH Terms: conditions — Sarcoma | interventions — apatinib; pirarubicin; Ifosfamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apatinib and Chemotherapy Test Group (Experimental): Apatinib 500mg, orally, once a day. One cycle every 4 weeks. Pirarubicin 75mg/m2 D1, intravenous infusion for 1-2 hours; every 4 weeks. Ifosfamide 2g/m2/d D1-D5, intravenously for 4-6 hours, 1 cycle every 4 weeks.
  Interventions: Drug: Apatinib Mesylate, Pirarubicin, Ifosfamide
- Apatinib Group (Active Comparator): Apatinib 500mg, orally, once a day. One cycle every 4 weeks.
  Interventions: Drug: Apatinib Mesylate
- Chemotherapy Group (Active Comparator): Pirarubicin 75mg/m2 D1, intravenous infusion for 1-2 hours; every 4 weeks. Ifosfamide 2g/m2/d D1-D5, intravenously for 4-6 hours, 1 cycle every 4 weeks.
  Interventions: Drug: Pirarubicin, Ifosfamide

INTERVENTIONS:
Drug: Apatinib Mesylate, Pirarubicin, Ifosfamide — Apatinib 500mg, orally, once a day. One cycle every 4 weeks. Pirarubicin 75mg/m2 D1, intravenous infusion for 1-2 hours; every 4 weeks. Ifosfamide 2g/m2/d D1-D5, intravenously for 4-6 hours, 1 cycle every 4 weeks.
  Arms: Apatinib and Chemotherapy Test Group
Drug: Apatinib Mesylate — Apatinib 500mg, orally, once a day. One cycle every 4 weeks.
  Arms: Apatinib Group
Drug: Pirarubicin, Ifosfamide — Pirarubicin 75mg/m2 D1, intravenous infusion for 1-2 hours; every 4 weeks. Ifosfamide 2g/m2/d D1-D5, intravenously for 4-6 hours, 1 cycle every 4 weeks
  Arms: Chemotherapy Group

SUMMARY:
To observe the efficacy of apatinib combined with AI regimen chemotherapy compared with AI regimen chemotherapy and single-agent apatinib in patients with unresectable soft tissue sarcoma. The main observations were progression-free survival (PFS) and progression-free control rate (PFR), followed by objective response rates (ORR, CR+PR), disease control rate (DCR, CR+PR+SD), and overall survival ( OS).

To observe the safety of apatinib combined with AI chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join the study, sign informed consent, and have good compliance;
2. A distantly metastatic or locally advanced and soft tissue sarcoma subject determined by the investigator not suitable for surgical treatment (Confirmed by pathology or cytology, except for gastrointestinal stromal tumors, cartilage-bone tumors, embryonic/acinar rhabdomyosarcoma, Ewing's sarcoma, and distant metastatic soft tissue tumors such as dermatofibrosarcoma And inflammatory myofibroblastic sarcoma, clear cell sarcoma and alveolar soft tissue sarcoma, etc).
3. The clinical staging is based on the TNM staging criteria of the American Joint Committee on Cancer Research (AJCC). At least one double-path measurable lesion according to CT or MR I;
4. Patients who have not previously received chemotherapy for soft-tissue sarcoma; or who have benefited from chemotherapy and who have relapsed or metastasized more than 6 months after discontinuation of the drug. The accumulated amount of anthracycline used in the past <450mg/m2.
5. 14~75 years old, PS score: 0~1 (Amputation patient can be relaxed to 2 points); the expected survival time is more than 3 months;
6. All acute toxic reactions caused by previous anti-tumor treatment or surgery are relieved to 0-1 before screening (according to NCI CTCAE version 4.03) or to the level specified by the enrollment/exclusion criteria (alopecia, etc. Except for toxicity that does not pose a safety risk to the subject);
7. There are sufficient organ and bone marrow functions, defined as follows: Blood routine (no blood transfusion within 14 days before treatment, no use of G-CSF, no use of drugs to correct), Neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L), Platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L), Hemoglobin (Hb) ≥ 9 g/dL (90 g/L); Blood chemistry, Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (Cockroft-Gault formula) ≥ 60 ml / min, Total bilirubin (TBIL) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 × ULN, liver metastases should be ≤ 5 × ULN; Coagulation, International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; Urine routine, Urine protein <2+; if urine protein ≥ 2+, 24-hour urine protein quantitation shows that the protein must be ≤ 1g; Thyroid function, Thyroid stimulating hormone (TSH) ≤ ULN; if abnormalities should be considered T3 and T4 levels, T3 and T4 levels can be selected;
8. Female subjects of childbearing age must undergo a serum pregnancy test within 7 days prior to treatment and the results are negative, and are willing to use a medically recognized effective contraceptive measure during the study period and within 3 months after the last administration of the study drug (eg: Intrauterine devices, contraceptives or condoms; for male subjects whose partners are women of childbearing age, surgical sterilization is required, or an effective method of contraception is recommended during the study period and within 3 months after the last study administration;
9. With my consent and signed informed consent, I am willing and able to follow planned visits, research treatments, laboratory tests and other testing procedures.

Exclusion Criteria:

1. The following treatments were received within 4 weeks of treatment: Radiotherapy, surgery, chemotherapy, immunization or molecular targeted therapy for tumors; Other clinical research drugs; Vaccination live attenuated vaccine;
2. Patients with previous chemotherapy failure or who have received anti-angiogenic targeted drugs within the past 3 months, such as Anlotinib, Pazopanib, Sorafenib, Sunitinib, Bevacizumab, Imatinib, Crizotinib, Apatinib, Regorafenib and Drugs such as endostatin;
3. Surgery and/or radiation therapy for soft tissue sarcomas is planned during the study (regardless of <5% of the bone marrow area);
4. Imaging diagnosis of central nervous system tumors;
5. Immune-suppressing drugs have been used within 14 days prior to initiation of treatment, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (That is, no more than 10 mg / day of prednisolone or equivalent physiological dose of other corticosteroids);
6. There is any active autoimmune disease or a history of autoimmune disease (Including but not limited to: Autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or asthma that have been completely relieved in childhood and currently do not require medical intervention may be included, or a history of allogeneic organ transplantation or a history of allogeneic hematopoietic stem cell transplantation);
7. Severe infections (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks prior to treatment, or unexplained fever >38.5 °C during screening/first administration;
8. High blood pressure, and excellent control without antihypertensive medication (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg);
9. There are significant clinically significant bleeding symptoms or clear bleeding tendency within 3 months before treatment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, vasculitis, etc. Or venous/venous thrombosis events occurring within 6 months prior to treatment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; or require long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥ 300 mg / day or clopidogrel ≥ 75 mg / day);
10. There were active heart disease in the 6 months before treatment, including myocardial infarction, severe/unstable angina. Echocardiography left ventricular ejection fraction <50%, poorly controlled arrhythmia (including QTcF interval men > 450 ms, women > 470 ms);
11. Any other malignant tumor was diagnosed within 3 years prior to treatment, except for adequately treated basal cells or squamous cell skin cancer or cervical carcinoma in situ;
12. It is known to be allergic to the study drug or any of its excipients;
13. Human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-positive and HBV DNA ≥ 500 IU/ml), Hepatitis C (positive hepatitis C antibody and higher detection limit of HCV-RNA than analytical methods);
14. At the discretion of the investigator, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, neurological or psychiatric disorders, etc.) that seriously compromise the safety of the subject, may confuse the findings, or affect the subject's completion of the study. Any other situation.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Within 2 years
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Disease control rate(DCR） | Within 2 years
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Objective tumor response rate(ORR) | Within 2 years
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Overall survival(OS) | Within 3 years
  OS is defined as the length of time from random assignment to death or to last contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital & Institute, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol